CLINICAL TRIAL: NCT06632795
Title: The Relationship Between Emotional Intelligence, Social Behavior, Sleep Quality and Academic Success in Students Studying in Health-Related Departments
Status: Not yet recruiting | Type: Observational
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Other Study IDs: Emotional Intelligence
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: University Students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to examine the relationships between emotional intelligence, positive social behavior, sleep quality, and academic achievement among students enrolled in health-related academic programs. Specifically, the study will investigate how emotional intelligence levels influence students' social behaviors and academic performance, while also assessing the role of sleep quality in these variables. Data will be collected using the Emotional Intelligence Scale, the Positive Social Behavior Scale, and the Epworth Sleepiness Scale. The findings of this study are expected to provide valuable insights into how emotional intelligence and sleep quality impact students' academic success and social behavior.

ELIGIBILITY:
Inclusion Criteria:

* Being a university student in health-related departments

Exclusion Criteria:

* Having any diagnosed physical or psychological illness

Ages: 17 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: University students studying health-related departments
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-21 (Estimated); Primary Completion 2024-12-09 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Emotional intelligence scale | Two months
  The scale is a 4-point Likert-type scale. The scale consists of 20 questions and four sub-dimensions (Well-being, Self-control, Emotionality and Sociability). A high score on the scale indicates that individuals have high levels of emotional intelligence.
Prosocial behavior scale | Two months
  It was used to measure prosocial behavioral tendencies among university students. The scale has five response options (1-Does not describe me at all, 5-Describes me very well).
Epworth sleepiness scale | Two months
  It questions the individual's general level of sleepiness. It aims to evaluate the chance of falling asleep or dozing off in eight different daily life situations (while sitting and reading a book, while watching television, while sitting quietly in a public place, while traveling in the car, while lying down in the afternoon, while talking to someone else, while sitting quietly after lunch without drinking alcohol, while in a car stopped for a few minutes in traffic).

SECONDARY OUTCOMES:
Academic Success Score | Two month
  Academic success scores of university students are examined.